CLINICAL TRIAL: NCT02253485
Title: Case-control Study of Antiviral Therapy During Entire and the Third Trimester of Pregnancy in Preventing MTCT of HBV in Mothers With High Serum HBV DNA Load
Brief Title: Efficacy of Antiviral Therapy in Pregnancy in Preventing Vertical Transmission of HBV in Mothers With a High Viral Load
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, The department of obstetrics and gynecology, Beijing Ditan Hospital
Other Study IDs: D121100003912001
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2012-08

CONDITIONS: Immune Globulin, Prophylaxis, Telbuvidine, Vaccine
Keywords: Mother-to-child transmission
MeSH Terms: interventions — Telbivudine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- telbivudine treated entire pregnancy: mothers in this group were treated with antiviral therapy during entire pregnancy for hepatitis, and their infants receive standard immunoprophylaxis for preventing MTCT of HBV.
  Interventions: Drug: telbivudine
- telbivudine treated in late pregnancy: mothers with high serum HBV DNA load were treated with antiviral therapy in late pregnancy, and their infants receive standard immunoprophylaxis for preventing MTCT of HBV.
  Interventions: Drug: telbivudine
- HBV DNA positive control: infants in this group born to mother with high serum HBV DNA load and receive standard immunoprophylaxis or additional HBIG injection at 1 month after birth for preventing MTCT of HBV.
- HBV DNA negative control: infants in this group born to a HBsAg positive and serum HBV DNA negative mothers and receive standard immunoprophylaxis for preventing MTCT of HBV

INTERVENTIONS:
Drug: telbivudine — in telbivudine treatment entire pregnancy group, mothers were treated with telbivudine during entire pregnancy for hepatitis B.
  in telbivudine treatment in late pregnancy group, mothers with high serum HBV DNA load receive telbivudine treatment in late pregnancy for preventing MTCT of HBV.
  Groups: telbivudine treated entire pregnancy; telbivudine treated in late pregnancy

SUMMARY:
Mother-to-child transmission (MTCT) is the most common route of hepatitis B virus (HBV) infection. After given standard immunoprophylaxis, MTCT still occurred in some infants born to a HBsAg positive mothers with high HBV DNA load. The main purpose of this study is evaluating the efficacy of methods used in blocking MTCT of HBV in infants born to a HBsAg positive mothers with high serum HBV DNA loads.

DETAILED DESCRIPTION:
This study contain 600 patients and compose groups as follow: (ⅰ) infants born to a HBsAg positive mothers with high HBV DNA load before delivery receive standard immunoprophylaxis( injection of HBIG 200IU at birth plus HBV vaccine at 0,1 and 6month); (ⅱ) infants born to a HBsAg positive mother with high HBV DNA load before delivery, and based on standard immunoprophylaxis receive addition injection of HBIG 200IU at 1 month after birth; (ⅲ) infants born to a HBsAg positive and high HBV DNA load mothers but treated with antiviral therapy in late pregnancy, receive standard immunoprophylaxis; (ⅳ) infants born to a HBsAg positive mothers treated with antiviral therapy during entire pregnancy for hepatitis receive standard immunoprophylaxis; (ⅴ) infants born to a HBsAg positive mother with serum HBV DNA negative receive standard immunoprophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* infants born to HBsAg positive mother HBsAg positive mother

Exclusion Criteria:

* mothers coinfected HIV or HCV

Max Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: this study would enroll 600 HBsAg positive mothers, including 240 cases with high serum HBV DNA load during pregnancy, 120 cases treated with antiviral therapy for hepatitis B, 120 cases with HBV DNA negative during pregnancy, 120 cases with high serum HBV DNA but receive antiviral therapy in late of pregnancy, and all of their infants.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
mother-to-child transmission of HBV | 7 months
  HBV infenction in infants at 7 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yi, Principal Investigator — Beijing Ditan Hospital

REFERENCES:
- [Derived] Yi W, Li MH, Xie Y, Wu J, Hu YH, Zhang D, Zhang Y, Cao WH. Prospective cohort study on the efficacy and safety of telbivudine used throughout pregnancy in blocking mother-to-child transmission of hepatitis B virus. J Viral Hepat. 2017 Nov;24 Suppl 1:49-56. doi: 10.1111/jvh.12788. PMID 29082650